CLINICAL TRIAL: NCT05219695
Title: Medical Imaging and Thermal Treatment for Breast Tumors Using Harmonic Motion Imaging (HMI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elisa Konofagou, Professor of Biomedical Engineering, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAS9859
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Fibroadenoma; Breast Cancer Stage I
MeSH Terms: conditions — Fibroadenoma; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMIgFUS (Experimental): Each study participants' tumors will be imaged using Harmonic Motion Imaging (HMI), an ultrasound elastography method. A central portion of the tumor will then be ablated and monitored using Harmonic Motion Imaging guided Focus Ultrasound (HMIgFUS). Only one portion of the tumor will be ablated; the other portions of the tumor, including tumor margins, will not be ablated. Following ablation, the tumor will be imaged again using HMI.
  Interventions: Procedure: Harmonic motion imaging guided focused ultrasound (HMIgFUS)

INTERVENTIONS:
Procedure: Harmonic motion imaging guided focused ultrasound (HMIgFUS) — Harmonic motion imaging guided focused ultrasound (HMIgFUS) is a combined treatment and imaging method, in which focused ultrasound (FUS) is used to thermally ablate tissue and harmonic motion imaging (HMI) is used for FUS guidance and monitoring. FUS applies high intensity focused ultrasound waves at its specified target to heat the tissue over a specified duration, causing cell death at the target area. HMI is an elasticity imaging technique which induces dynamic tissue vibrations at the target for tissue elasticity characterization.
  One of the inclusion criteria for this study is that participants must be scheduled for surgical excision of their breast tumor. In this study, HMIgFUS will be applied to anesthetized participants immediately prior to their scheduled surgery. HMI imaging will also be performed immediately prior to and after HMIgFUS application.

SUMMARY:
The objective of this study is to demonstrate the initial clinical feasibility of using Harmonic Motion Imaging (HMI) for Focused Ultrasound Surgery (FUS) guidance and monitoring in patients with benign and stage 1 non-metastatic breast cancers. The investigators hypothesize that changes in HMI parameters will inform progression of FUS ablation.

DETAILED DESCRIPTION:
Patients with small solid tumors without positive lymph nodes have the highest survival rate. However, especially for patients with benign tumors (most common in younger women) and older patients (>65 years old) who fit these criteria, an alternative treatment technique that is less invasive than the current surgical or invasive ablative intervention may be more beneficial. FUS is a noninvasive, non-ionizing treatment procedure that precisely focuses and delivers a large amount of ultrasound energy to the target area, causing localized temperature rise and cell necrosis at the target. The main advantage of focused ultrasound ablation (FUS) is that it avoids surgery. Without surgery, recovery from the procedure is much faster, patients may experience less pain, and cosmetological results may be improved.

The efficacy and safety of FUS rely heavily on treatment monitoring. Treatment imaging techniques currently used include MRI and ultrasound Bmode imaging. Magnetic resonance imaging (MRI) thermometry is used to detect the temperature rise across the FUS treatment area. However, MRI guidance can be expensive and time-consuming compared to ultrasound-based HIFU guidance methods. Conventional B-mode based 'hyperecho' tracking can be challenging for HIFU monitoring, as it is sensitive to cavitation, which occurs at high temperatures.

HMI is an ultrasound elasticity method that can provide measurements of the locally generated mechanical response and inherent mechanical properties of tissues . The result is a new image that contains unique localized information on the relative stiffness in and around the tumor. The investigators have shown in pre-clinical data that HMI has the ability to monitor mechanical changes in tissue that occur with ablation. The combination of FUS with HMI monitoring is termed HMI guided FUS, or HMIgFUS.

This study aims to evaluate the HMI technique for monitoring FUS ablation in a clinical setting. Eligible and consenting patients will be imaged using HMI, and then will undergo HMIgFUS at a central position inside the tumor. The tumor will be imaged using HMI again following ablation. Following our study, the patients will undergo their scheduled surgery. The purpose of this study is to evaluate HMIgFUS in a lower risk setting, as the tumor will be excised following our study, to better inform future studies, in which surgery may not be needed.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥18
* Patients with fibroadenoma (benign tumor) or early-stage, non-metastatic breast cancer (stage I without the involvement of axillary lymph nodes)
* Scheduled to receive surgical resection of the tumor by the clinical care team (ideal target lesion upper boundary should be deeper than 1 cm below the skin, and the ideal size of the lesion should be 2-5 cm in diameter)

Exclusion Criteria:

* Pregnant or lactating women
* Patients with breast implants
* Patients with a history of laser or radiation therapy to the targeted breast
* Patients who have received or are scheduled to receive thermal ablation or treatment of the tumor (other than surgery) as part of clinical care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with ablation | From the date of ablation and imaging to the date of pathological results (approximately 1 week)
  To identify markers of ablation progression using HMIgFUS images, thereby predicting whether ablation occurred or not. The investigators will also use differences in HMI imaging performed before and after ablation to assess the presence of ablation. The results from both of these methods will be validated with pathological findings, to determine whether ablation was achieved.
R2 value of ablated lesion depth | From the date of ablation and imaging to the date of pathological results (approximately 1 week)
  The depth of the lesion (in mm away from the surface of the skin) as shown on HMIgFUS images will be compared and validated with pathological findings.
R2 value of ablated lesion width | From the date of ablation and imaging to the date of pathological results (approximately 1 week)
  The width of the lesion (in mm laterally across the lesion) as shown on HMIgFUS images will be compared and validated with pathological findings.
R2 value of ablated lesion area | From the date of ablation and imaging to the date of pathological results (approximately 1 week)
  The area of the lesion (in mm^2) as shown on HMIgFUS images will be compared and validated with pathological findings.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Konofagou, PhD, Principal Investigator — Professor of Biomedical Engineering
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers.

REFERENCES:
- [Background] Han Y, Wang S, Payen T, Konofagou E. Fast lesion mapping during HIFU treatment using harmonic motion imaging guided focused ultrasound (HMIgFUS) in vitro and in vivo. Phys Med Biol. 2017 Apr 21;62(8):3111-3123. doi: 10.1088/1361-6560/aa6024. Epub 2017 Mar 21. PMID 28323638
- [Background] Han Y, Wang S, Hibshoosh H, Taback B, Konofagou E. Tumor characterization and treatment monitoring of postsurgical human breast specimens using harmonic motion imaging (HMI). Breast Cancer Res. 2016 May 9;18(1):46. doi: 10.1186/s13058-016-0707-3. PMID 27160778